CLINICAL TRIAL: NCT01289119
Title: An International, Multicenter, Randomized, Double-blind, Placebo-controlled, Phase 3 Study to Determine the Efficacy and Safety of SYR-322 When Used in Subjects With Type 2 Diabetes
Brief Title: Efficacy and Safety of Alogliptin in Participants With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYR-322_02; U1111-1118-3681 (Registry Identifier: WHO); SYR-322_308 (Other: Takeda ID)
Record Dates: First submitted 2011-02-01; First posted 2011-02-03 (Estimated); Results first posted 2013-03-22 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 Diabetes Mellitus; Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — alogliptin; Metformin; Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Placebo (Placebo Comparator): Participants received alogliptin placebo-matching tablets, orally once daily for up to 16 weeks.
  Interventions: Drug: Placebo to alogliptin
- Alogliptin Monotherapy (Experimental): Participants received alogliptin 25 mg tablets, orally, once daily for up to 16 weeks.
  Interventions: Drug: Alogliptin
- Metformin (Other): Participants continued to receive their stable dose of metformin (≥1000 mg/day) and also received alogliptin placebo-matching tablets, orally once daily for up to 16 weeks.
  Interventions: Drug: Placebo to alogliptin; Drug: Metformin
- Metformin + Alogliptin Add-on Therapy (Experimental): Participants continued to receive their stable dose of metformin (≥1000 mg/day) and also received alogliptin 25 mg tablets, orally, once daily for up to 16 weeks.
  Interventions: Drug: Alogliptin; Drug: Metformin
- Pioglitazone (Other): Participants continued to receive their stable dose of pioglitazone with or without metformin, and also received alogliptin placebo-matching tablets, orally once daily for up to 16 weeks.
  Interventions: Drug: Placebo to alogliptin; Drug: Pioglitazone
- Pioglitazone + Alogliptin Add-on Therapy (Experimental): Participants continued to receive their stable dose of pioglitazone with or without metformin and also received alogliptin, 25 mg tablets orally once daily for up to 16 weeks.
  Interventions: Drug: Alogliptin; Drug: Pioglitazone

INTERVENTIONS:
Drug: Alogliptin — Alogliptin tablets
  Other Names: SYR-322
  Arms: Alogliptin Monotherapy; Metformin + Alogliptin Add-on Therapy; Pioglitazone + Alogliptin Add-on Therapy
Drug: Placebo to alogliptin — Alogliptin placebo-matching tablets.
  Arms: Metformin; Pioglitazone; Placebo
Drug: Metformin — Stable metformin dose
  Other Names: Fortamet; Glucophage; Glumetza
  Arms: Metformin; Metformin + Alogliptin Add-on Therapy
Drug: Pioglitazone — Stable pioglitazone dose
  Other Names: Actos
  Arms: Pioglitazone; Pioglitazone + Alogliptin Add-on Therapy

SUMMARY:
The purpose of the study is to determine the efficacy of alogliptin compared to placebo when given alone or as add-on therapy to metformin or add-on to pioglitazone (with or without metformin).

DETAILED DESCRIPTION:
Diabetes is a chronic illness associated with microvascular complications such as nephropathy (kidney disease), retinopathy (eye damage) and neuropathy (nervous system damage). Diabetes is also associated with macrovascular complications including cardiovascular disease (heart disease), stroke and peripheral vascular disease (narrowing or blockage of blood vessels). These complications are associated with reduced quality of life and increased morbidity and mortality.

Takeda is developing SYR-322 (alogliptin) for improvement of glycemic control in patients with Type 2 diabetes mellitus.

Evaluations of alogliptin and its clinical efficacy have been conducted in multiple countries including the United States and Japan. This study will be conducted as a multi-center clinical trial in order to validate the efficacy and safety of alogliptin on type 2 diabetes population within Asia.

Participants who qualified for the study were stratified into 1 of the 3 therapy groups based upon their background antidiabetic therapy before being randomized 1:1 to receive either alogliptin 25 mg once daily or matching placebo once daily.

* Monotherapy group - patients who had been treated with diet and exercise for at least 2 months prior to screening.
* Add-on to metformin therapy group - patients who had been treated with metformin for at least 3 months and at a stable dose (≥1000 mg/day) for at least 8 weeks prior to screening.
* Add-on to pioglitazone therapy group - patients who had been treated with a stable dose of pioglitazone alone or in combination with metformin at a stable dose for at least 8 weeks prior to screening.

ELIGIBILITY:
Inclusion Criteria:

* Has a historical diagnosis of Type 2 Diabetes Mellitus.
* Has a body mass index between acceptable range.
* Is experiencing inadequate glycemic control.
* Body weight keeps constant.
* Females of childbearing potential and males who are sexually active agree to use routinely adequate contraception from signing of informed consent throughout the duration of the study and for 30 days after last dose.

Exclusion Criteria:

* Has participated in another clinical study within the past 90 days or has received any investigational compound within 30 days prior to randomization.
* Has a systolic blood pressure beyond the acceptable range at Screening visit.
* Has New York Heart Association Class III or IV heart failure regardless of therapy.
* Has any major illness or debility that in the investigator's opinion prohibits the subject from completing the study.
* Has a history of hypersensitivity or allergies to any DPP-4 inhibitor.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 506 (Actual)
Dates: Start 2010-12; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Professor Study Chair, Study Chair — Takeda
Locations (21):
- China (19):
  - Beijing, Beijing Municipality
  - Fuzhou, Fujian
  - Xiamen, Fujian
  - Guangzhou, Guangdong
  - Haikou, Hainan
  - Harbin, Heilongjiang
  - Jingzhou, Hubei
  - Shiyan, Hubei
  - Changsha, Hunan
  - Wuxi, Jiangsu
  - Nanchang, Jiangxi
  - Changchun, Jilin
  - Shenyang, Liaoning
  - Jinan, Shandong
  - Shanghai, Shanghai Municipality
  - Xi’an, Shanxi
  - Tianjin, Tianjin Municipality
  - Kunming, Yunnan
  - Hangzhou, Zhejiang
- Hong Kong, Hong Kong, Hong Kong
- Taipei County, Taiwan

REFERENCES:
- [Derived] El-Damanawi R, Stanley IK, Staatz C, Pascoe EM, Craig JC, Johnson DW, Mallett AJ, Hawley CM, Milanzi E, Hiemstra TF, Viecelli AK. Metformin for preventing the progression of chronic kidney disease. Cochrane Database Syst Rev. 2024 Jun 4;6(6):CD013414. doi: 10.1002/14651858.CD013414.pub2. PMID 38837240

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 30 investigative sites in China, Taiwan province and Hong Kong from 23 December 2010 to 19 December 2011.
Pre-assignment Details: Participants with a historical diagnosis of Type 2 diabetes mellitus who were experiencing inadequate glycemic control were stratified into 1 of the 3 therapy groups based upon their background antidiabetic therapy before being randomized 1:1 to receive either alogliptin 25 mg once daily or matching placebo once daily.
Groups:
- Pioglitazone: Participants continued to receive their stable dose of pioglitazone with or without metformin and also received alogliptin placebo-matching tablets, orally once daily for up to 16 weeks.
Period: Overall Study
Arm/Group | Placebo | Alogliptin Monotherapy | Metformin | Metformin + Alogliptin Add-on Therapy | Pioglitazone | Pioglitazone + Alogliptin Add-on Therapy
Started | 93 | 92 | 98 | 99 | 63 | 61
Treated | 92 (Patients who took at least one dose of double-blind study drug.) | 92 | 98 | 99 | 63 | 61
Completed | 84 | 83 | 89 | 93 | 58 | 57
Not Completed | 9 | 9 | 9 | 6 | 5 | 4
Not completed — Adverse Event | 2 | 1 | 0 | 2 | 1 | 0
Not completed — Major Protocol Deviation | 2 | 1 | 3 | 0 | 2 | 1
Not completed — Lost to Follow-up | 0 | 3 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 4 | 2 | 4 | 3 | 1 | 1
Not completed — Pregnancy | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 1 | 1 | 1 | 1 | 1
Not completed — Other | 1 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Alogliptin Monotherapy | Metformin | Metformin + Alogliptin Add-on Therapy | Pioglitazone | Pioglitazone + Alogliptin Add-on Therapy | Total
Number analyzed (Participants) | 93 | 92 | 98 | 99 | 63 | 61 | 506
Age Continuous [Mean (Standard Deviation); unit: years] | 53.1 (8.88) | 51.6 (10.41) | 53.2 (9.46) | 53.0 (9.88) | 51.8 (10.37) | 52.6 (9.44) | 52.6 (9.71)
Age, Customized [Number; unit: participants]
  <65 Years | 81 | 80 | 86 | 85 | 56 | 52 | 440
  ≥65 years | 12 | 12 | 12 | 14 | 7 | 9 | 66
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 37 | 50 | 48 | 24 | 33 | 231
  Male | 54 | 55 | 48 | 51 | 39 | 28 | 275
Race/Ethnicity, Customized [Number; unit: participants] | 93 | 92 | 98 | 99 | 63 | 61 | 506
Region of Enrollment [Number; unit: participants]
  Taiwan | 1 | 0 | 2 | 3 | 0 | 0 | 6
  Hong Kong | 1 | 2 | 2 | 4 | 0 | 0 | 9
  China | 91 | 90 | 94 | 92 | 63 | 61 | 491
Height [Mean (Standard Deviation); unit: cm] | 165.4 (7.19) | 165.9 (8.61) | 164.8 (8.47) | 165.7 (9.06) | 166.2 (8.87) | 163.0 (7.06) | 165.2 (8.31)
Weight [Mean (Standard Deviation); unit: kg] | 70.86 (10.464) | 71.16 (11.065) | 69.67 (11.792) | 71.20 (13.473) | 72.44 (11.989) | 67.59 (11.989) | 70.55 (11.856)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 25.86 (3.002) | 25.79 (3.086) | 25.54 (2.876) | 25.75 (3.122) | 26.13 (3.031) | 25.32 (3.223) | 25.73 (3.042)
Diabetes duration [Mean (Standard Deviation); unit: years] | 2.12 (2.845) | 1.86 (2.369) | 5.33 (3.873) | 5.38 (4.335) | 4.85 (4.724) | 5.80 (5.300) | 4.11 (4.215)
HbA1c [Number; unit: participants]
  <8.0% | 47 | 48 | 54 | 55 | 34 | 32 | 270
  ≥8.0% | 46 | 44 | 44 | 44 | 29 | 29 | 236
Stable Daily Dose of Metformin [Mean (Standard Deviation); unit: mg] — Participant population for this measure for each treatment arm: 0, 0, 98, 99, 50, 50; Total population: 297
  mg | NA (NA) — Participants in this arm were not taking Metformin | NA (NA) — Participants in this arm were not taking Metformin | 1484.2 (451.09) | 1472.2 (417.31) | 1355.0 (431.80) | 1295.0 (506.82) | 1426.6 (450.90)
Stable Daily Dose of Pioglitazone [Mean (Standard Deviation); unit: mg] — Participant population for this measure for each treatment arm: 0, 0, 0, 0, 63, 61; Total population: 124
  mg | NA (NA) — Participants in this arm were not taking Pioglitazone | NA (NA) — Participants in this arm were not taking Pioglitazone | NA (NA) — Participants in this arm were not taking Pioglitazone | NA (NA) — Participants in this arm were not taking Pioglitazone | 21.9 (11.37) | 20.2 (7.19) | 21.0 (9.55)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c)
Description: The change from Baseline in HbA1c (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at Week 16. Least squares means are derived from an analysis of covariance (ANCOVA) model with treatment as a fixed effect, and baseline HbA1c as a covariate for the monotherapy, baseline HbA1c with baseline metformin dose as covariates for the metformin therapy, baseline HbA1c with baseline metformin therapy status and baseline pioglitazone dose as covariates for the pioglitazone therapy.
Time Frame: Baseline and Week 16.
Population: The full analysis set, consisting of all patients who received at least one dose of double-blind study drug and who had a baseline assessment and at least one post-baseline HbA1c assessment. Last observation carried forward was utilized.
Measure: Least Squares Mean (Standard Error); unit: percentage glycosylated hemoglobin
Arm/Group | Placebo | Alogliptin Monotherapy | Metformin | Metformin + Alogliptin Add-on Therapy | Pioglitazone | Pioglitazone + Alogliptin Add-on Therapy
Number analyzed (Participants) | 90 | 90 | 97 | 98 | 63 | 60
percentage glycosylated hemoglobin | -0.42 (0.074) | -0.99 (0.074) | -0.22 (0.065) | -0.91 (0.065) | -0.25 (0.097) | -0.76 (0.101)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin Monotherapy; The analysis was conducted at the 2-sided 5% significance level without a multiplicity adjustment; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA model with treatment as a fixed effect, and baseline HbA1c as a covariate; LS Mean Difference = -0.58, 95% CI 2-sided [-0.78 to -0.37]
Statistical Analysis 2: Comparison: Metformin vs Metformin + Alogliptin Add-on Therapy; The analysis was conducted at the 2-sided 5% significance level without a multiplicity adjustment; Test type: Superiority or Other; p < 0.001, ANCOVA — ANCOVA model with treatment as a fixed effect, and baseline HbA1c with baseline metformin dose as covariates; LS Mean Difference = -0.69, 95% CI 2-sided [-0.87 to -0.51]
Statistical Analysis 3: Comparison: Pioglitazone vs Pioglitazone + Alogliptin Add-on Therapy; The analysis was conducted at the 2-sided 5% significance level without a multiplicity adjustment; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA model with treatment as a fixed effect, and baseline HbA1c with baseline metformin therapy status and baseline pioglitazone dose as covariates; LS Mean Difference = -0.52, 95% CI 2-sided [-0.75 to -0.28]

2. Secondary Outcome: Change From Baseline in HbA1c Over Time
Description: The change from Baseline in HbA1c (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) at Weeks 4, 8 and 12. Least squares means are derived from an analysis of covariance (ANCOVA) model with treatment as a fixed effect, and baseline HbA1c as a covariate for the monotherapy, baseline HbA1c with baseline metformin dose as covariates for the metformin therapy, baseline HbA1c with baseline metformin therapy status and baseline pioglitazone dose as covariates for the pioglitazone therapy.
Time Frame: Baseline and Weeks 4, 8 and 12.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage glycosylated hemoglobin
Arm/Group | Placebo | Alogliptin Monotherapy | Metformin | Metformin + Alogliptin Add-on Therapy | Pioglitazone | Pioglitazone + Alogliptin Add-on Therapy
Number analyzed (Participants) | 92 | 92 | 98 | 99 | 63 | 61
percentage glycosylated hemoglobin
  Week 4 (n=90, 88, 97, 98, 63, 60) | -0.24 (0.059) | -0.56 (0.059) | -0.15 (0.036) | -0.43 (0.036) | -0.09 (0.064) | -0.44 (0.066)
  Week 8 (n=90, 90, 97, 98, 63, 60) | -0.39 (0.068) | -0.86 (0.068) | -0.15 (0.057) | -0.66 (0.057) | -0.31 (0.094) | -0.70 (0.098)
  Week 12 (n=90, 90, 97, 98, 63, 60) | -0.41 (0.078) | -0.99 (0.078) | -0.24 (0.069) | -0.86 (0.068) | -0.25 (0.102) | -0.77 (0.106)

3. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose Over Time
Description: The change from Baseline in fasting plasma glucose (FPG) at Weeks 4, 8, 12 and 16. Least squares means are derived from an ANCOVA model with treatment as a fixed effect, and baseline FPG as a covariate for the monotherapy, baseline FPG with baseline metformin dose as covariates for the metformin therapy, baseline FPG with baseline metformin therapy status and baseline pioglitazone dose as covariates for the pioglitazone therapy.
Time Frame: Baseline and Weeks 4, 8, 12 and 16.
Population: The full analysis set, consisting of all patients who received at least one dose of double-blind study drug and who had a baseline assessment and at least one post-baseline FPG assessment. Last observation carried forward was utilized.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo | Alogliptin Monotherapy | Metformin | Metformin + Alogliptin Add-on Therapy | Pioglitazone | Pioglitazone + Alogliptin Add-on Therapy
Number analyzed (Participants) | 92 | 92 | 98 | 99 | 63 | 61
mmol/L
  Week 4 (n=89, 87, 97, 97, 63, 60) | -0.331 (0.1221) | -0.719 (0.1235) | -0.251 (0.1454) | -0.985 (0.1454) | 0.284 (0.2505) | -0.985 (0.2603)
  Week 8 (n=89, 89, 97, 97, 63, 60) | -0.330 (0.1224) | -1.015 (0.1224) | -0.235 (0.1397) | -1.265 (0.1397) | -0.038 (0.2503) | -0.924 (0.2600)
  Week 12 (n=89, 89, 97, 97, 63, 60) | -0.411 (0.1515) | -1.123 (0.1515) | -0.335 (0.1600) | -1.270 (0.1600) | -0.187 (0.2484) | -1.177 (0.2581)
  Week 16 (n=89, 89, 97, 97, 63, 60) | -0.317 (0.1556) | -1.243 (0.1556) | -0.512 (0.1565) | -1.240 (0.1565) | -0.114 (0.2579) | -1.070 (0.2679)

4. Secondary Outcome: Percentage of Participants With Marked Hyperglycemia
Description: Marked Hyperglycemia was defined as fasting plasma glucose greater than or equal to 200 mg/dL (11.1 mmol/L).
Time Frame: Randomization to Week 16.
Population: The full analysis set, consisting of all patients who received at least one dose of double-blind study drug and who had a baseline assessment and at least one post-baseline assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Alogliptin Monotherapy | Metformin | Metformin + Alogliptin Add-on Therapy | Pioglitazone | Pioglitazone + Alogliptin Add-on Therapy
Number analyzed (Participants) | 89 | 89 | 97 | 97 | 63 | 60
percentage of participants | 16.9 | 4.5 | 25.8 | 13.4 | 23.8 | 8.3

5. Secondary Outcome: Change From Baseline in Body Weight
Description: The change between body weight measured at Baseline and body weight measured at Weeks 8 and 16. The least squares means are derived from an ANCOVA model with treatment as a fixed effect, and baseline body weight as a covariate for the monotherapy, baseline body weight with baseline metformin dose as covariates for the add-on to metformin therapy, baseline body weight with baseline metformin therapy status and baseline pioglitazone dose as covariates for the add-on to pioglitazone therapy.
Time Frame: Baseline and Weeks 8 and 16.
Population: The full analysis set, consisting of all patients who received at least one dose of double-blind study drug and who had a baseline assessment and at least one post-baseline weight assessment. Last observation carried forward was utilized.
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Placebo | Alogliptin Monotherapy | Metformin | Metformin + Alogliptin Add-on Therapy | Pioglitazone | Pioglitazone + Alogliptin Add-on Therapy
Number analyzed (Participants) | 92 | 92 | 98 | 99 | 63 | 61
kg
  Week 8 (n=87, 86, 94, 96, 63, 59) | -1.04 (0.210) | -0.71 (0.211) | -0.82 (0.170) | -0.43 (0.168) | -0.74 (0.286) | -0.15 (0.304)
  Week 16 (n=88, 87, 94, 96, 63, 59) | -1.55 (0.244) | -0.89 (0.245) | -1.06 (0.219) | -0.76 (0.217) | -0.68 (0.364) | -0.10 (0.388)

6. Secondary Outcome: Percentage of Participants With HbA1c ≤6.5% at Week 16
Description: Clinical response was assessed by the percentage of participants with HbA1c (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) less than or equal to 6.5% at Week 16.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Alogliptin Monotherapy | Metformin | Metformin + Alogliptin Add-on Therapy | Pioglitazone | Pioglitazone + Alogliptin Add-on Therapy
Number analyzed (Participants) | 90 | 90 | 97 | 98 | 63 | 60
percentage of participants | 12.2 | 36.7 | 4.1 | 21.4 | 9.5 | 30.0

7. Secondary Outcome: Percentage of Participants With HbA1c ≤7.0% at Week 16
Description: Clinical response was assessed by the percentage of participants with HbA1c (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) less than or equal to 7.0% at Week 16.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Alogliptin Monotherapy | Metformin | Metformin + Alogliptin Add-on Therapy | Pioglitazone | Pioglitazone + Alogliptin Add-on Therapy
Number analyzed (Participants) | 90 | 90 | 97 | 98 | 63 | 60
percentage of participants | 30.0 | 63.3 | 25.8 | 55.1 | 31.7 | 61.7

8. Secondary Outcome: Percentage of Participants With HbA1c ≤7.5% at Week 16
Description: Clinical response was assessed by the percentage of participants with HbA1c (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) less than or equal to 7.5% at Week 16.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Alogliptin Monotherapy | Metformin | Metformin + Alogliptin Add-on Therapy | Pioglitazone | Pioglitazone + Alogliptin Add-on Therapy
Number analyzed (Participants) | 90 | 90 | 97 | 98 | 63 | 60
percentage of participants | 53.3 | 81.1 | 50.5 | 80.6 | 47.6 | 85.0

9. Secondary Outcome: Percentage of Participants With a Decrease in HbA1c ≥ 0.5%
Description: Clinical response was assessed by the percentage of participants with a decrease from Baseline in HbA1c of greater than or equal to 0.5% at Week 16.
Time Frame: Baseline and Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Alogliptin Monotherapy | Metformin | Metformin + Alogliptin Add-on Therapy | Pioglitazone | Pioglitazone + Alogliptin Add-on Therapy
Number analyzed (Participants) | 90 | 90 | 97 | 98 | 63 | 60
percentage of participants | 41.1 | 84.4 | 37.1 | 70.4 | 42.9 | 76.7

10. Secondary Outcome: Percentage of Participants With a Decrease in HbA1c ≥1.0%
Description: Clinical response was assessed by the percentage of participants with a decrease from Baseline in HbA1c of greater than or equal to 1.0% at Week 16.
Time Frame: Baseline and Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Alogliptin Monotherapy | Metformin | Metformin + Alogliptin Add-on Therapy | Pioglitazone | Pioglitazone + Alogliptin Add-on Therapy
Number analyzed (Participants) | 90 | 90 | 97 | 98 | 63 | 60
percentage of participants | 20.0 | 50.0 | 9.3 | 45.9 | 19.0 | 46.7

11. Secondary Outcome: Percentage of Participants With a Decrease in HbA1c ≥1.5%
Description: Clinical response was assessed by the percentage of participants with a decrease from Baseline in HbA1c of greater than or equal to 1.5% at Week 16.
Time Frame: Baseline and Week 16.
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Alogliptin Monotherapy | Metformin | Metformin + Alogliptin Add-on Therapy | Pioglitazone | Pioglitazone + Alogliptin Add-on Therapy
Number analyzed (Participants) | 90 | 90 | 97 | 98 | 63 | 60
percentage of participants | 7.8 | 23.3 | 1.0 | 22.4 | 7.9 | 8.3

12. Secondary Outcome: Percentage of Participants With a Decrease in HbA1c ≥2.0%
Description: Clinical response was assessed by the percentage of participants with a decrease from Baseline in HbA1c of greater than or equal to 2.0% at Week 16.
Time Frame: Baseline and Week 16.
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Alogliptin Monotherapy | Metformin | Metformin + Alogliptin Add-on Therapy | Pioglitazone | Pioglitazone + Alogliptin Add-on Therapy
Number analyzed (Participants) | 90 | 90 | 97 | 98 | 63 | 60
percentage of participants | 2.2 | 8.9 | 0.0 | 9.2 | 1.6 | 3.3

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAE) were defined as any adverse events that started on or after the date of the first dose of double-blind study drug and within 14 days after the date of the last dose of double-blind study drug.
Description: The investigator had to document any occurrence of adverse events at each visit, and the occurrence of abnormal laboratory findings at applicable visits. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Placebo | Alogliptin Monotherapy | Metformin | Metformin + Alogliptin Add-on Therapy | Pioglitazone | Pioglitazone + Alogliptin Add-on Therapy
Serious Adverse Events (participants affected / at risk) | 2/92 | 2/92 | 3/98 | 0/99 | 0/63 | 1/61
Other Adverse Events (participants affected / at risk) | 11/92 | 12/92 | 8/98 | 7/99 | 14/63 | 18/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=92) | Alogliptin Monotherapy (N=92) | Metformin (N=98) | Metformin + Alogliptin Add-on Therapy (N=99) | Pioglitazone (N=63) | Pioglitazone + Alogliptin Add-on Therapy (N=61)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cholangitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Intraductal papilloma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Lacunar infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=92) | Alogliptin Monotherapy (N=92) | Metformin (N=98) | Metformin + Alogliptin Add-on Therapy (N=99) | Pioglitazone (N=63) | Pioglitazone + Alogliptin Add-on Therapy (N=61)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 6 | 0 | 0 | 4 | 13
Upper respiratory tract infection (Infections and infestations) | 3 | 5 | 5 | 3 | 6 | 2
Urinary tract infection (Infections and infestations) | 6 | 2 | 2 | 2 | 1 | 4
Blood triglycerides increased (Investigations) | 1 | 2 | 2 | 2 | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.